CLINICAL TRIAL: NCT00114257
Title: A Phase I Study of 5-AZA-2'-Deoxycytidine and Depsipeptide in Patients With Relapsed/Refractory Leukemia, Myelodysplastic Syndromes, or Myeloproliferative Disease
Brief Title: Decitabine and FR901228 in Treating Patients With Relapsed or Refractory Leukemia, Myelodysplastic Syndromes, or Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02657; MDA-2004-0674; NCI-5563; CDR0000433040 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute promyelocytic leukemia (M3); relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; chronic myelomonocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; Philadelphia chromosome negative chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute basophilic leukemia; adult acute eosinophilic leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute | interventions — Decitabine; romidepsin

ARMS (1):
- Arm I (Experimental): Patients receive decitabine IV over 1 hour on days 1-5 and 8-12 and FR901228 (depsipeptide) IV over 4 hours on days 5 and 12 OR days 5, 12, and 19. Treatment repeats every 4-6 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing complete remission for 1 year are removed from the study.
  Cohorts of 6 patients receive escalating doses of decitabine and FR901228 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: decitabine; Drug: romidepsin

INTERVENTIONS:
Drug: decitabine
Drug: romidepsin

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine and FR901228 in treating patients with relapsed or refractory leukemia, myelodysplastic syndromes or myeloproliferative disorders. Drugs used in chemotherapy, such as decitabine and FR901228, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. FR901228 may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer. Giving decitabine together with FR901228 may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose and recommended phase II dose of decitabine and FR901228 (depsipeptide) in patients with relapsed or refractory leukemia, myelodysplastic syndromes, or myeloproliferative disease.

II. Determine the safety and tolerability of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive decitabine IV over 1 hour on days 1-5 and 8-12 and FR901228 (depsipeptide) IV over 4 hours on days 5 and 12 OR days 5, 12, and 19. Treatment repeats every 4-6 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing complete remission for 1 year are removed from the study.

Cohorts of 6 patients receive escalating doses of decitabine and FR901228 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia

    * Previously untreated patients > 60 years of age who are not eligible for front-line therapy are eligible for this study
  * Acute lymphoblastic leukemia
  * Chronic myelogenous leukemia (CML)

    * Documented hematologic resistance to imatinib mesylate OR no cytogenetic response after 12 months of prior treatment with imatinib mesylate
    * Philadelphia chromosome-negative CML allowed provided disease is resistant to standard therapy (e.g., hydroxyurea) OR disease progressed (blasts > 5% and platelet count < 100,000/mm^3) during standard therapy
  * Myelodysplastic syndromes

    * International Prognostic Scoring System risk category ≥ intermediate-1
    * Patients who are not eligible for front-line therapy are eligible for this study
  * Myeloproliferative disease
  * Chronic lymphocytic leukemia

    * Failed or progressed during ≥ 1 prior fludarabine-based therapy AND alemtuzmab
  * Acute promyelocytic leukemia

    * Progressed after prior treatment with standard chemotherapy, tretinoin, and arsenic trioxide
  * Chronic myelomonocytic leukemia

    * Resistant to standard therapy (e.g., hydroxyurea) OR disease progressed (blasts > 5% and platelet count < 100,000/mm^3) during standard therapy
* Relapsed or refractory disease
* No known brain or meningeal disease

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* More than 8 weeks

Hepatic

* Bilirubin < 2 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine < 2 mg/dL

Cardiovascular

* QTc < 500 msec
* LVEF > 40% by MUGA
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No uncontrolled angina
* No left ventricular hypertrophy by EKG
* No history of serious ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No other significant cardiac disease

Immunologic

* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to study drugs
* No ongoing or active infection
* No HIV positivity

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Chemotherapy

* Recovered from prior chemotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) unless there is evidence of rapidly progressive disease

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Other

* No concurrent agents that cause QTc prolongation
* No other concurrent investigational or commercial agents or therapies for the malignancy
* No concurrent hydrochlorothiazide

  * Concurrent potassium-conserving combinations (e.g., Maxide® or Dyazide®) or other antihypertensive agents allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Toxicity at 6 weeks after each course

SECONDARY OUTCOMES:
Complete and partial response at 6 weeks after each course

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Issa, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States